CLINICAL TRIAL: NCT02819245
Title: Impact of Age on Surgical Outcome of Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Hongda Bao, Resident and research scientist, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-01-15-scoliosis
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Age before and after 18 years old (Other): Surgical treatment before and after skeletal maturity
  Interventions: Procedure: posterior correction and fusion

INTERVENTIONS:
Procedure: posterior correction and fusion

SUMMARY:
This is a study prospectively enrolling adolescent idiopathic scoliosis (AIS) patients and try to find how the age will impact the surgical outcome of AIS.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent idiopathic scoliosis patients; undergoing posterior correction surgery; with minimum 5 years follow-up; with full-spine radiography.

Exclusion Criteria:

* with spinal tumor; with hip disease; without quality of life measurements.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of coronal Cobb angle | From immediate post-operative until at least 10 years follow-up
  Cobb angles, including thoracic and lumbar Cobb angle, are measured from coronal radiographs with validated software (Surgimap).

SECONDARY OUTCOMES:
Improvement of sagittal profile | From immediate post-operative until at least 10 years follow-up
  Sagittal profile, described sagittal radiographic parameters such as thoracic kyphosis and lumbar lordosis, is measured with validated software (Surgimap).
Health-related quality of life (HRQOL) | From immediate post-operative until at least 10 years follow-up
  HRQOL measurements include Short Form 36 (SF-36), Scoliosis Research Society (SRS) 22 questionnaire and Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Yong Qiu, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No